CLINICAL TRIAL: NCT02866604
Title: Comparison of an Isotonic Balanced Fluid, Sterofundin® , With 0.9% Saline in Traumatic Brain Injury(TBI)
Acronym: FLUID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201510-1766
Record Dates: First submitted 2016-05-23; First posted 2016-08-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Brain Injuries
Keywords: Traumatic brain injury; isotonic balanced fluid
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic | interventions — sterofundin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strerofundin (Active Comparator): Days of intervention: 3 days
  Interventions: Procedure: Sterofundin
- 0.9% saline (Active Comparator): Days of intervention: 3 days
  Interventions: Procedure: 0.9% saline

INTERVENTIONS:
Procedure: Sterofundin
  Arms: Strerofundin
Procedure: 0.9% saline
  Arms: 0.9% saline

SUMMARY:
The main objective of this study is to compare the clinical outcomes of TBI patients receiving only Sterofundin or 0.9% saline as main fluid therapy.

DETAILED DESCRIPTION:
Study Design: Prospective single centre double-blind randomized controlled trial

Study endpoints/outcomes

Primary outcomes:

* 30 day mortality
* Functional neurological outcomes at 6 months based on Extended Glasgow Outcome Scale (GOS-E)

Secondary outcomes:

* Acid-base and electrolyte balance
* Daily mean change in intracranial pressure (ICP)
* Episodes of intracranial hypertension
* Duration of mechanical ventilation
* Length of ICU stay and ICU mortality

Study Duration: 2 years Site: UMMC. Departments involved: Emergency Medicine, Surgery, Anaesthesiology and Pharmacy

Methodology. Investigators will assess patients admitted to the Emergency Department, UMMC, for eligibility.

Randomisation:

Investigators will randomize patients in a 1:1 ratio to either 0.9% saline intravenous fluid group or Sterofundin® intravenous fluid group. An independent statistician not involved with the research will perform a block of eight randomisation using computerised number generator list.

Conduct of study The Department of Pharmacy will identically seal all 0.9% saline and Sterofundin® intravenous fluid bottles and label them, according to their type, as either A or B. The patients, investigators and medical and nursing staff will not be aware of the designation of the letters A and B to the fluids.

Investigators will administer the study fluid will immediately after patient randomisation and this will last for 72 hours.

Other general care of the traumatic brain injury patients from both study arms will continue as per Neurosurgical Unit protocol and Brain Trauma Foundation guidelines.

Data handling

Investigators will collect all data relevant to both primary and secondary outcomes (see also attached proforma):

Statistical analysis Investigators will conduct students t test, Chi squared and the Mann-Whitney U test as appropriate. Investigators will adjust results with univariable and multivariable logistic regression and report their odds ratio. Investigators will present survival analysis using Kaplan Meier curves and compare them using log rank test.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 and 65 years of age
* Non-penetrating moderate (GCS 9-12) or severe (GCS 3-8) traumatic brain injury
* Within 12 hours since the recorded time of injury

Exclusion Criteria:

* Pregnancy
* Polytrauma
* Cardiac arrest at presentation
* GCS of three with bilateral fixed dilated pupils,
* Evidence of severe cardiac, respiratory, renal or liver dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
30 day mortality | 30 days
Functional neurological outcomes at 6 months based on Extended Glasgow Outcome Scale (GOS-E) | 180 days

SECONDARY OUTCOMES:
Acid-base balance | 3 days
  through out intervention period
Daily mean change in intracranial pressure (ICP) | 3 days
  through out intervention period
Episodes of intracranial hypertension | 3 days
  through out intervention period
Duration of mechanical ventilation | 3 days
  through out intervention period
Length of ICU stay | 30 days
  through out intervention period
electrolyte balance | 3 days
ICU mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaya Medical Centre, Petaling Jaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No